CLINICAL TRIAL: NCT05051163
Title: A Randomized Trial to Investigate Strategies to Reduce Mortality Among HIV-infected and HIV-exposed Children Admitted With Severe Acute Malnutrition in Mulago Hospital, Kampala, Uganda
Brief Title: Strategies to Reduce Mortality Among HIV-infected and HIV-exposed Children Admitted With Severe Acute Malnutrition
Acronym: REDMOTHIV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Associate Professor, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC.REF.2020-165; HS1277ES (Other: Uganda National Council For Science and Technology)
Record Dates: First submitted 2021-08-06; First posted 2021-09-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: HIV-1-infection; Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Ceftriaxone; Ampicillin; Gentamicins

STUDY DESIGN:
Intervention Model Description: Open label parallel group randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftriaxone (Experimental): Ceftriaxone will be administered intravenously at a dose of 50 - 75mg/kg once daily
  Interventions: Drug: Ceftriaxone Sodium
- Ampicillin and Gentamicin (Active Comparator): 1. Ampicillin will be administered intravenously at a dose of 50mg/kg 6hourly
  2. Gentamicin will be administered intravenously at a dose 5mg/kg once daily
  Interventions: Drug: Ampicillin; Drug: Gentamicin

INTERVENTIONS:
Drug: Ceftriaxone Sodium — 7 days of once daily dosing
  Other Names: ZEFONE-1000
  Arms: Ceftriaxone
Drug: Ampicillin — 7 days of 6 hourly dosing
  Other Names: AMPIMAX-500
  Arms: Ampicillin and Gentamicin
Drug: Gentamicin — 7 days of once daily dosing
  Other Names: GENTAMICIN INJECTION
  Arms: Ampicillin and Gentamicin

SUMMARY:
This study to investigate whether empiric use of an antibiotic with greater antimicrobial sensitivity (ceftriaxone) than standard-of-care (ampicillin plus gentamicin) will reduce mortality among HIV-infected/HEU children admitted to Mwanamugimu Nutrition Unit, Mulago Hospital, Kampala, Uganda.

DETAILED DESCRIPTION:
Background

HIV-infected and HIV-exposed-uninfected children (HEU) are at increased risk of developing malnutrition. Severely malnourished children have high mortality rates, but mortality is higher in those that are HIV-infected. Preliminary audits at the Mwanamugimu Nutrition Unit, Mulago Hospital, in 2014 showed that 43% of the severely malnourished children that died were HIV-infected/HEU, despite only 30% of admissions being HIV-infected/HEU, with deaths due to infections in 90% of cases.

Objectives

This study aims to investigate whether empiric use of an antibiotic with greater antimicrobial sensitivity (ceftriaxone) than standard-of-care (ampicillin plus gentamicin) will reduce mortality among HIV-infected/HEU children admitted to Mwanamugimu Nutrition Unit. Secondary objectives include: comparing length of hospitalization, weight-for-height, weight-for-age and height-for-age z-scores between ceftriaxone versus standard of care (ampicillin and gentamicin) treatment arms; ascertaining the pattern/antimicrobial sensitivity of pathogens among participants; determining the prevalence and factors associated with HIV-infection among severely malnourished children; and evaluating the pharmacokinetics (PK) of lopinavir/ritonavir (LPV/r) among severely malnourished HIV-infected children.

Methods

This will be an open label randomized controlled trial involving 300 children; 76 HIV-infected (current mortality - 33%) and 224 HEU (current mortality - 26%). The participants will be randomized to receive 1week of ceftriaxone (n= 150) or standard-of-care (ampicillin/gentamicin) (n=150), in addition to other routine care; the ratio of HIV-infected to HEU (1:3) in this sample is reflective of the current proportions of the HIV-infected and HEU children admitted at Mwanamugimu Nutrition Unit. The trial's primary outcome will be in hospital mortality. 300 randomised children provides >80% power to detect reductions in mortality from the expected 28% to 14%, allowing for 10% noncompliance/lost-to-follow-up in each group. Secondary outcomes will be: length of hospitalization; weight-for-height, weight-for-age and height-for-age z-scores; and pattern/antimicrobial sensitivity of pathogens. In addition, 280 severely malnourished children of unknown serostatus will be tested for HIV at admission to determine the prevalence and factors associated with HIV-infection. 280 children provide 80% power to determine the prevalence of HIV-infection. Furthermore, all the HIV-infected children on LPV/r will each provide sparse pharmacokinetic (PK) samples to evaluate the PK of LPV/r among malnourished children. In this PK sub-study, geometric means of steady-state LPV PK parameters [Area Under the Curve (AUC) 0-12h, maximum concentration (Cmax) and concentration at 12 hours after dose (C12h)] will be determined. The PK parameters (AUC 0-12h, Cmax, C12) will then be put in pharmacokinetic-pharmacodynamic (PK-PD) models to determine optimal doses for the study population.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected children aged 1 to 59 months admitted at Mwanamugimu Nutrition Unit with severe acute malnutrition
2. HIV exposed but uninfected children aged 1 to 59 months admitted at Mwanamugimu Nutrition Unit with severe acute malnutrition
3. For prevalence of HIV-infection sub-study, children presenting with severe acute malnutrition on admission at Mwanamugimu Nutrition Unit.
4. For PK sub-study, the child should have been on antiretroviral therapy for at least 2weeks and should have been in hospital for at least 2weeks.

Exclusion Criteria:

* For PK sub-study; a child with documented poor adherence to antiretroviral therapy.
* For PK sub-study; a child known to have vomited the drug on the sampling day.

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-06-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | 4 weeks
  Cumulative incidence

SECONDARY OUTCOMES:
Length of hospitalization | 90 days
  Number of days
Weight-for-height z-score | 90 days
  Change from baseline
Weight-for-age z-score | 90 days
  Change from baseline
Height-for-age z-score | 90 days
  Change from baseline
Pattern and antimicrobial sensitivity of pathogens | 7 days
  Frequency
HIV infection | Baseline
  Prevalence
Area under the curve (AUC 0- 12h) | 12hours
  Geometric means
Maximum concentration (Cmax) | 12hours
  Geometric means
Concentration at 12hours post dose (C12h) | 12hours
  Geometric means

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University College of Health Sciences, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: Yes
When results are required as part of a meta-analysis or as secondary data.
Supporting Information: Study Protocol
Time Frame: 1 year after end of data collection
Access Criteria: On request to Principal Investigator

REFERENCES:
- [Derived] Musiime V, Kiggwe A, Beinomugisha J, Kakooza L, Thembo-Mwesige J, Nkinzi S, Naguti E, Atuhaire L, Segawa I, Ssengooba W, Mukonzo JK, Babirekere-Iriso E, Musoke P. Strategies to Reduce Mortality Among Children Living With HIV and Children Exposed to HIV but Are Uninfected, Admitted With Severe Acute Malnutrition at Mulago Hospital, Uganda (REDMOTHIV): A Mixed Methods Study. Front Pediatr. 2022 Jun 24;10:880355. doi: 10.3389/fped.2022.880355. eCollection 2022. PMID 35813373